CLINICAL TRIAL: NCT07050693
Title: Efficacy of A 2'-Fucosylactose-based Food Supplement on the Prevention of Respiratory and Gastrointestinal Infections in Schhol-attended Children: a Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: Efficacy of a 2'-Fucosylactose-based Food Supplement on the Prevention of Respiratory and Gastrointestinal Infections.
Acronym: IMMUNOSICK24
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Professor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IMMUNOSICK24
Record Dates: First submitted 2025-03-21; First posted 2025-07-03 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Gastroenteric Tract; Respiratory Tract; Infections; Gastroenteric Infections
Keywords: food supplement; gastroenteric infection
MeSH Terms: conditions — Infections | interventions — Vitamins; Zinc

STUDY DESIGN:
Intervention Model Description: Randomized double bind with placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Nobody knows the randomization code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): 50 children will take the product under study based on Vitamin D, Zinc, Beta glucan, 2'Fucosyllactose
  Interventions: Dietary Supplement: Vitamin + Zinc + micronutrient mixture
- Placebo (Placebo Comparator): 50 children will take a carbohydrate-based control product (maltodextrin)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin + Zinc + micronutrient mixture — a dietary supplement containing Vitamin D, Zinc, Beta glucan WELLMUNE WGP, 2'Fucosyllactose.
  Other Names: Experimental arm
  Arms: Experimental
Dietary Supplement: Placebo — Placebo is identical to intervention product
  Arms: Placebo

SUMMARY:
Respiratory and gastrointestinal infections are frequent problems in children under 4 years of age, especially after the start of schooling. These conditions are facilitated by an incomplete maturation of the immune system and by the anatomical and functional structure of the respiratory and gastrointestinal tract still in development.

Functional foods derived from the fermentation of cow's milk with probiotic strains have been proposed for the prevention of infectious diseases in children. Several products have been investigated, sometimes with conflicting results. Some scientific evidence has shown that the administration of Vitamin D, Zinc, Beta glucan, 2'-Fucosyllactose can stimulate the immune defenses and reduce the number and severity of infectious episodes. In particular, 2'-fucosyllactose is one of the oligosaccharides of breast milk. It has both a prebiotic and immunoregulatory action since it is able to prevent the adhesion of pathogens to epithelial surfaces and subsequent translocation.

Healthy school-going children aged between 12 and 48 months, who attend school at least 5 days a week, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy school-going children aged 12 to 48 months who attend school at least 5 days a week

Exclusion Criteria:

* Age less than 12 months and more than 48 months;
* Concomitant presence of chronic diseases
* Congenital heart disease;
* Tuberculosis;
* Functional gastrointestinal disorders;
* Gastrointestinal or urinary surgery of the respiratory tract;
* Autoimmune diseases;
* Immunodeficiencies;
* Chronic inflammatory bowel diseases;
* Celiac disease;
* Cystic fibrosis;
* Metabolic diseases;
* Lactose intolerance;
* Tumors;
* Chronic lung diseases and malformations of the gastrointestinal tract;
* Food allergies;
* Eosinophilic esophagitis;
* Other hypereosinophilic diseases of the gastrointestinal tract;
* Diarrhea at enrollment;
* Severe malnutrition (z score for weight/height less than 3SD);
* Taking antibiotics and/or pre/pro/symbiotics/immunostimulants within 2 weeks of starting the study;
* Breastfeeding in progress

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | The dietary supplement and placebo will be administered for three months from the date of enrollment.
  The primary aim of the study will be the percentage of children who will present at least one infectious episode (acute gastroenteritis, rhinitis, otitis, pharyngitis, laryngitis, tracheitis) diagnosed by the pediatrician during the 3-month study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatria Trambusti, Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siziba LP, Mank M, Stahl B, Kurz D, Gonsalves J, Blijenberg B, Rothenbacher D, Genuneit J. Associations of Human Milk Oligosaccharides With Otitis Media and Lower and Upper Respiratory Tract Infections up to 2 Years: The Ulm SPATZ Health Study. Front Nutr. 2021 Oct 25;8:761129. doi: 10.3389/fnut.2021.761129. eCollection 2021. PMID 34760912
- [Background] Etzold S, Bode L. Glycan-dependent viral infection in infants and the role of human milk oligosaccharides. Curr Opin Virol. 2014 Aug;7:101-7. doi: 10.1016/j.coviro.2014.06.005. Epub 2014 Jul 19. PMID 25047751
- [Background] Hatakka K, Savilahti E, Ponka A, Meurman JH, Poussa T, Nase L, Saxelin M, Korpela R. Effect of long term consumption of probiotic milk on infections in children attending day care centres: double blind, randomised trial. BMJ. 2001 Jun 2;322(7298):1327. doi: 10.1136/bmj.322.7298.1327. PMID 11387176